CLINICAL TRIAL: NCT04236180
Title: Specialised Paediatric Palliative Care: Assessing Family, Healthcare Professionals and Health System Outcomes in a Multi-site Context of Various Care Settings
Brief Title: Effectiveness of Specialised Paediatric Palliative Care
Acronym: SPhAERA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: University of Basel (Other); Cantonal Hospital of Aarau, Switzerland (Other); University Children's Hospital Basel (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-INV-001
Record Dates: First submitted 2019-03-15; First posted 2020-01-22 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Paediatric Palliative Care
Keywords: Paediatrics; Palliative Care

STUDY DESIGN:
Intervention Model Description: Interventional multi-centre study with a hybrid design to determine the clinical effectiveness (comparative effectiveness research) of an existing SPPC programme, while gathering information on its delivery and potential implementation in a real-life situation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): Patients enrolled in the Specialised Paediatric Palliative Care (SPPC) programme at the University Children's Hospital Zurich.
  Interventions: Other: Specialised Paediatric Palliative Care (SPPC)
- Comparison Group (No Intervention): Patients treated at the Children's Hospital Aarau, University Children's Hospital Basel, and the University Hospital Inselspital Bern.

INTERVENTIONS:
Other: Specialised Paediatric Palliative Care (SPPC) — All services provided to children/families by a member of the multiprofessional SPPC team in Zurich according to local guidelines will be considered as study intervention. This includes direct consultation of the patient/family, as well as patient-/family-related consultation of the frontline care team. Bereavement support is considered an integrated part of SPPC and after the death of a child, follow-up bereavement support is routinely offered at the individual or group level as appropriate for parents and siblings.
  Arms: Intervention Group

SUMMARY:
This study evaluates the effectiveness of an existing Specialised Paediatric Palliative Care programme and reports on its potential to improve patient-, family-, health professionals-, and healthcare-related outcomes. Data will be compared between an intervention and a comparison group.

DETAILED DESCRIPTION:
The number of children and adolescents living with life-limiting conditions and potentially in need for specialised paediatric palliative care (SPPC) is rising. As a highly complex subfield of palliative care, paediatric palliative care focuses on the support and involvement of the entire family, and on the impact not only at the patient level, but also at the family and health systems level. Ideally, a specialised multiprofessional team fills the complex healthcare needs of children and their families. A consultative care model might be well-suited to address each family's most important needs. The question, however, of how SPPC is beneficial for whom and under what circumstances remain largely unanswered as validation of innovative care programmes in controlled studies is lacking.

This study's overall target is to evaluate the effectiveness of SPPC and to report on its potential to improve patient-, family-, health professional-, and healthcare-related outcomes. The primary objective is to explore how SPPC influences the quality of life (QOL) of caregivers, i.e. parents. Secondary objectives are to explore how SPPC influences the QOL of patients including their symptom severity and distress as well as the QOL of their siblings and of healthcare professionals not specialised in PPC. Further objectives are to determine whether the provision of SPPC reduces the utilisation of healthcare resources and direct and indirect health-related costs for families, and to evaluate implementation outcomes such as adoption, i.e., the uptake of SPPC.

This interventional multi-centre study will apply a hybrid design to determine the clinical effectiveness (comparative effectiveness research) of an existing SPPC programme, while gathering information on its delivery and potential implementation in a real-life situation.

This study will be conducted in compliance with the protocol, the current version of the Declaration of Helsinki, the ICH-GCP as well as all national legal and regulatory requirements.

ELIGIBILITY:
Children suffering from a life-limiting condition and potentially in need of SPPC, their parents and siblings as applicable will be eligible to enter the study, along with all HCP involved in their care at all study sites. The potential need for SPPC is defined per indication criteria based on the Zurich SPPC programme's guidelines:

* Increase in (unplanned) hospital admissions during the last months
* Medical adverse events from which the child is not recovering completelyIncreasing symptom burden
* Unsatisfactory response to treatments
* Conflicting treatment goals
* Estimated life expectancy less than 6-12 months
* Patient's/parents' wish for PC support

Inclusion criteria:

* Children, aged 0-18 years, suffering from a life-limiting condition of various origins and potentially in need of SPPC (for Zurich, additionally enrolment in the SPPC programme)
* Parents (mothers and fathers) of included children
* Siblings, aged >8 years, of included families
* All health care professionals involved in the care of included families
* Proficiency in French or German language
* Signed Informed Consent after being informed

Exclusion criteria:

* Neonates with medical complications due to prematurity and/or birth complications and treated in a neonatal intensive care unit
* Children with an estimated life expectancy of <48 hours

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Caregiver QOL - QOLLTI-F Questionnaire | Up to day 330 after study entry
  Longitudinal assessment of self-reported caregiver (parental) Quality of Life (QOL) using the QOLLTI-F (Quality of Life in Life Threatening Illness - Family Carer Version) questionnaire.

SECONDARY OUTCOMES:
Change in Child's QOL - DISABKIDS Chronic Generic Measure (DCGM-37) Questionnaire | Up to day 330 after study entry
  Longitudinal assessment of child's Quality of Life using the DCGM-37 DISABKIDS questionnaire.
Change in child's symptoms - Memorial Symptom Assessment Scale (MSAS) Questionnaire | Up to day 330 after study entry
  Longitudinal assessment of child's symptoms by using the Memorial Symptom Assessment Scale (MSAS) questionnaire. MSAS assesses severity, frequency and distress for symptom evaluation using separate 4 or 5 point Likert scales. Higher values are associated with higher symptom burden.
Change in Siblings QOL - KIDSSCREEN-27 Questionnaire | Up to day 630 after study entry
  Longitudinal assessment of sibling's health related Quality of Life using the KIDSSCREEN-27 questionnaire.
Professional's QOL (ProQOL) Questionnaire | Cross-sectional at the end of study year 1
  Assessing self-reported healthcare professional's Quality of Life using the ProQOL questionnaire.
Professional's QOL (ProQOL) Questionnaire | Cross-sectional at the end of study year 2
  Assessing self-reported healthcare professional's Quality of Life using the ProQOL questionnaire.
Chang in grief - "Würzburger Trauerinventar (WüTi)" Questionnaire | Up to 1 year after the child's death
  Longitudinal assessment of parental grief processes using the "Würzburger Trauerinventar (WüTi)" questionnaire.
Change in parental QOL during bereavement - WHOQOL-BREF Questionnaire | Up to 1 year after the child's death
  Longitudinal assessment of parental Quality of Life during bereavement using the WHO Quality of Life-BREF questionnaire.

OTHER OUTCOMES:
Number of hospital admissions as assessed longitudinally via chart review | Up to day 330 after study entry
  Number of admissions including number of emergency and/or outpatient consultations and number of admissions to a pediatric palliative care unit. Routine data, chart review, longitudinally during the child's palliative care phase.
Number of resuscitations | Up to day 330 after study entry
  Routine data, chart review, continuously during the child's palliative care phase.
Number of invasive procedures | Up to day 330 after study entry
  E.g. surgery and imaging requiring sedation. Routine data, chart review, continuously during the child's palliative care phase.
Length of Stay (LOS) | Up to day 330 after study entry
  Total length of hospital stay per admission. Routine data, chart review, continuously during the child's palliative care phase.
Number of days receiving professional community home care services | Up to day 330 after study entry
  Routine data, chart review, continuously during the child's palliative care phase.
Place of Death | Place of death will be recorded, if the patient dies within 1 year after study enrollment.
  (Hospital, Home, Hospice, Other) Data extraction from routine data/cart reviews at time of death.
Effective costs charged and paid for by formal payers | Up to day 630 after study entry
  Cost estimations based on resource utilization combined with publicly available sources or retrieved from payers for each family who consented.
Family household expenditures | after 1 year or at child's death; 1 year after the child's death
  Direct and indirect household expenditures. Household data obtained using questionnaires.
SPPC - Paediatric Palliative Screening Scale (PaPas-Scale) Questionnaire | For each patient at baseline (study enrollment), through study completion, ca. 2 years.
  Identification of patients in need of specialised paediatric palliative care using the Paediatric Palliative Screening Scale (PaPas-Scale) questionnaire. Higher scores indicate a higher need for paediatric palliative care.
Sense of coherence (SOC) Questionnaire | For each family at baseline (study enrollment), through study completion, ca. 2 years.
  Assessment of self-reported Family Sense of Coherence with the FSOC questionnaire.
Family hardiness (FH) Questionnaire | For each family at baseline (study enrollment), through study completion, ca. 2 years.
  Assessing the internal strengths and cooperativeness, the resourcefulness and willingness to learn and the sense of having control over life circumstances by using the Family Hardiness Index (FHI) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Zimmermann, PhD RN, Principal Investigator — University Children's Hospital, Zurich
Locations (4):
- Switzerland (4):
  - Cantonal Children's Hospital, Aarau
  - University Children's Hospital, Basel
  - Department of Pediatrics, University Hospital Inselspital, Bern
  - University Children's Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mitterer S, Zimmermann K, Fink G, Simon M, Gerber AK, Bergstrasser E. Hospitalization- and death-related financial and employment effects in parents of children with life-limiting conditions: a fixed-effects analysis. Eur J Pediatr. 2024 Oct;183(10):4215-4227. doi: 10.1007/s00431-024-05680-7. Epub 2024 Jul 10. PMID 38985175
- [Derived] Gerber AK, Feuz U, Zimmermann K, Mitterer S, Simon M, von der Weid N, Bergstrasser E. Work-related quality of life in professionals involved in pediatric palliative care: a repeated cross-sectional comparative effectiveness study. Palliat Care Soc Pract. 2024 May 9;18:26323524241247857. doi: 10.1177/26323524241247857. eCollection 2024. PMID 38737405
- [Derived] Zimmermann K, Simon M, Scheinemann K, Tinner Oehler EM, Widler M, Keller S, Fink G, Mitterer S, Gerber AK, von Felten S, Bergstraesser E. Specialised Paediatric PAlliativE CaRe: Assessing family, healthcare professionals and health system outcomes in a multi-site context of various care settings: SPhAERA study protocol. BMC Palliat Care. 2022 Nov 2;21(1):188. doi: 10.1186/s12904-022-01089-x. PMID 36324132